CLINICAL TRIAL: NCT01326585
Title: Effect of Dexamethasone on Postoperative Symptoms of Scleral Buckling Surgery Patients: a Randomized Control Trial
Brief Title: Study Trial of Dexamethasone Use for Alleviation of Symptoms After Scleral Buckle Eye Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Toronto (Other)
Responsible Party: Dr. Mark Mandelcorn, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 0911-A
Record Dates: First submitted 2011-03-28; First posted 2011-03-31 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2011-01

CONDITIONS: Retinal Detachment
Keywords: Scleral Buckling; Dexamethasone; Post-operative Nausea and Vomiting
MeSH Terms: conditions — Retinal Detachment; Vomiting | interventions — dexamethasone 21-phosphate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Dexamethasone (Experimental): Subjects receive intravenous intraoperative dexamethasone
  Interventions: Drug: Dexamethasone Sodium Phosphate Injection
- Saline solution (Placebo Comparator): Subjects receive intravenous intraoperative normal saline solution
  Interventions: Drug: Saline Injection

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate Injection — 8mg (2cc of 4mg/mL solution), IV solution, 1-time dose during surgery
  Arms: Dexamethasone
Drug: Saline Injection — 2cc of 0.9% normal saline, IV injection, 1-time dose during surgery
  Arms: Saline solution

SUMMARY:
Dexamethasone is a medication that has been shown to have clear anti-nausea, anti-inflammatory, and painkilling properties. Dexamethasone is currently used to manage postoperative symptoms of a variety of surgical procedures. However, its effect has not been validated for scleral buckling surgery, which is used to treat retinal detachment, a medical emergency that can lead to permanent blindness. In this study, the investigators will randomly administer dexamethasone to half of scleral buckling surgery patients, and a placebo to the other half. The investigators will then compare the postoperative symptoms of the two groups in order to determine whether dexamethasone should be used for scleral buckling surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-79 years old
* Scheduled for scleral buckle surgery to treat a retinal detachment
* Consent to participate in study

Exclusion Criteria:

* Pregnant or nursing
* Prior treatment with steroids
* Severe diabetes mellitus (HbA1c > 8%)
* Use of opioids, sedatives, or any kind of analgesics <1 week before scleral buckling surgery
* History of alcohol or drug abuse

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Subjective Level of Postoperative Nausea | At 1 and 7 days post-surgery
  Assessed through patient survey, measured by 10cm visual analogue scale
Subjective Level of Postoperative Pain | 1 and 7 days post-surgery
  Assessed by patient survey, measured by Wong-Baker FACES Pain Rating Scale

SECONDARY OUTCOMES:
Subjective rating of post-operative lid edema | At 1 and 7 days post-surgery
  Assessed by investigator, rated "mild", "moderate", or "severe"
Subjective rating of postoperative chemosis | 1 and 7 days post-surgery
  Assessed by investigator, recorded as "mild", "moderate", or "severe"

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mandelcorn, MD FRCSC, Principal Investigator — University Health Network, Toronto; Rajeev Muni, MD FRCSC, Principal Investigator — Unity Health Toronto; Daniel B Rootman, MSc MD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario